CLINICAL TRIAL: NCT03254810
Title: A Phase 1 Randomized Blinded Single Dose Comparison of the Safety and Pharmacokinetics of SYN060 Compared to Adalimumab (Humira®) From North American and European Sources in Healthy Adult Subjects
Brief Title: Comparison of the Safety and PK of SYN060 to Humira® in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synermore Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYN060-001
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SYN060 (Experimental): a single 0.57 mg/kg dose of SYN060
  Interventions: Biological: SYN060
- Adalimumab North American source (Active Comparator): a single 0.57 mg/kg dose of adalimumab from North American source
  Interventions: Biological: Adalimumab North American source
- Adalimumab European source (Active Comparator): a single 0.57 mg/kg dose of adalimumab from European source
  Interventions: Biological: Adalimumab European source

INTERVENTIONS:
Biological: SYN060 — a single subcutaneous 0.57 mg/kg dose of SYN060
  Arms: SYN060
Biological: Adalimumab North American source — a single subcutaneous 0.57 mg/kg dose of adalimumab (Humira®) reference product from North American source
  Arms: Adalimumab North American source
Biological: Adalimumab European source — a single subcutaneous 0.57 mg/kg dose of adalimumab (Humira®) reference product from European source
  Arms: Adalimumab European source

SUMMARY:
This is a single site, parallel randomized, double blinded comparison of the safety, pharmacokinetics, and immunogenicity of a single 0.57 mg/kg dose of SYN060 to a single 0.57 mg/kg dose of adalimumab (Humira®) reference product from North American and European sources. The study is open to healthy individuals on no medications that might confound the results of this safety study.

DETAILED DESCRIPTION:
This is a single site, parallel randomized, double blinded comparison of the safety, pharmacokinetics, and immunogenicity of a single 0.57 mg/kg dose of SYN060 to a single 0.57 mg/kg dose of adalimumab (Humira®) reference product from North American and European sources. The study is open to healthy individuals on no medications that might confound the results of this safety study.

A total of 90 subjects will be randomized in a 1:1:1 ratio to from a centrally generated randomization schedule to SYN060 or adalimumab of American or European sources resulting in 30 subjects in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 50 years of age, inclusive
2. Body mass index between 18 and 30 kg/m², inclusive
3. Female subjects physically capable of pregnancy (i.e., not sterilized and still menstruating or within 1 year of the last menses if menopausal) must:

   1. Agree to avoid pregnancy from the Study Day screening visit through six months after receipt of Study Drug.
   2. If in a sexual relationship with a man, use an acceptable method of avoiding pregnancy during this period, still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring or intrauterine device (IUD).
4. Women of childbearing potential must have a negative serum pregnancy test within 24 hours preceding receipt of the dose.
5. Can understand and sign the informed consent document, can communicate with the investigator and provide updated contact information as needed for the duration of the study, has no current plans to move from the study area for the duration of the study, and can understand and comply with the requirements of the protocol.

Exclusion Criteria:

1. Acute illness on Study Day 1
2. Oral temperature ≥37.5°C on Study Day 1
3. Inability to discontinue daily medications other than oral contraceptives or other hormonal therapy.
4. Receipt of an immunoglobulin or blood product within 90 days prior to Study Day 1
5. Any receipt of adalimumab, or other licensed monoclonal antibody
6. Any receipt of another investigational product within 4 weeks or 4 half-lives whichever is longer prior to Study Day 1
7. Abnormal laboratory values per local laboratory parameters from blood collected at screening prior to Study Day 1 randomization as follows:

   * Severe anemia, defined as haemoglobin <100 g/L or hematocrit <0.3 L/L
   * absolute neutrophil count, below lower limit of normal (LLN)
   * white blood cell count above upper limit of normal (ULN) or below LLN (i.e., must be within normal limits)
   * ALT, AST, alkaline phosphatase (ALP) above ULN with exception that a one of the three values may be permitted up to 10% above ULN.
   * Creatinine above upper limit of normal ,
   * INR, or activated partial thromboplastin time (APTT) above ULN
8. Abnormal screening urinalysis result that is, per the investigator, clinically significant, or a screening urine dipstick result of ≥2+ protein
9. Positive screening urine test for illicit drugs (amphetamines, methamphetamines, barbiturates, benzodiazepine, cocaine, opiates, PCP, MDMA, methadone)
10. History of systemic allergic reactions, to more than one medication.
11. History or evidence of malignancy.
12. Receipt of immunosuppressive medications other than inhaled or topical immunosuppressant drugs such as corticosteroids within 45 days prior to Study Day 1
13. Hepatitis B surface antigen positive, HIV positive, hepatitis C antibody positive
14. Uncontrolled Type 2 Diabetes or Type I diabetes
15. History systemic fungal infection.
16. Shared a residence within the last year with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis
17. Previous medical history that may compromise the safety of the subject in the study, including but not limited to: severe impairment of pulmonary function or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease or poorly controlled epilepsy
18. History or evidence on physical examination of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety of the Study Drug
19. History or evidence of tuberculosis infection
20. Positive Quantiferon test
21. Chest X ray with evidence of malignancy or chronic infection (such as tuberculosis or other)
22. Any current medical, psychiatric, occupational, or substance abuse problem such as alcoholism that, in the opinion of the investigator, will make it unlikely that the subject will comply with the protocol.
23. Elective surgery that would interfere with participation.
24. Live virus vaccination within 60 days and during the study.
25. Blood donation less than 30 days prior to Study Day 1.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
AUC0-last (area under the concentration-time curve from time zero to the last non-zero concentration) and AUC0-inf (area under the concentration-time curve from time zero to infinity) | 85 days
  AUC0-last and AUC0-inf will be estimated using non-compartmental analysis fpr SYN060 to adalimumab (Humira®) from North American and European sources.
Cmax (maximum observed concentration) | 85 days
  Cmax will be estimated using non-compartmental analysis for SYN060 and adalimumab (Humira®) from North American and European sources
Residual area (%AUCextrap) [percent extrapolated area under the curve to infinity calculated as 100*(1- AUC0-last / AUC0-inf)] | 85 days
  Residual area (%AUCextrap) will be estimated using non-compartmental analysis for SYN060 and adalimumab (Humira®) from North American and European sources
Tmax (time of observed Cmax) | 85 days
  Tmax will be estimated using non-compartmental analysis for SYN060 and adalimumab (Humira®) from North American and European sources
t½ (elimination half-life) | 85 days
  t½ will be estimated using non-compartmental analysis for SYN060 and adalimumab (Humira®) from North American and European sources
λz (elimination rate constant) | 85 days
  λz will be estimated using non-compartmental analysis for SYN060 and adalimumab (Humira®) from North American and European sources
CL/F (apparent body clearance, calculated as Dose/AUC0-inf) | 85 days
  CL/F will be estimated using non-compartmental analysis for SYN060 and adalimumab (Humira®) from North American and European sources
Vz/F [apparent volume of distribution, calculated as Dose/ (λz x AUC0-inf)] | 85 days
  Vz/F will be estimated using non-compartmental analysis for SYN060 and adalimumab (Humira®) from North American and European sources

SECONDARY OUTCOMES:
Adverse event incidence of SYN060 compared to adalimumab (Humira®) from North American and European sources | 85 days
  Safety monitoring will include vital signs (blood pressure, temperature, pulse, oximetry and respiration rates), physical examination, electrocardiogram (ECG) and clinical laboratory tests (serum chemistry, hematology, troponins, creatinine phosphokinase [CPK], human anti-SYN060 antibodies, human anti-adalimumab antibodies and urinalysis). Adverse events will be recorded throughout the study and will be coded using the most current version of MedDRA (Medical Dictionary for Regulatory Activities) at the time of study commencement.
anti-SYN060 antibodies | 85 days
  The development of anti-SYN060 antibodieswill be determined on Study Days 0, and 7 through 85, or the last blood specimen available for subjects who leave the study prior to Day 85. The development of anti-SYN060 antibodies will be analyzed as a continuous measure across categorical groups and compared to anti-adalimumab antibodies with descriptive statistics.
anti-adalimumab antibodies | 85 days
  The development of anti-adalimumab antibodies will be determined on Study Days 0, and 7 through 85, or the last blood specimen available for subjects who leave the study prior to Day 85. The development of anti-adalimumab antibodies will be analyzed as a continuous measure across categorical groups and compared to anti-SYN060 antibodies with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Niquita Tugiono, MD, Principal Investigator — Nucleus Network, Center for Clinical Studies Study Site
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No